CLINICAL TRIAL: NCT06840366
Title: Effectiveness of a Motor Rehabilitation Program and Its Impact on Functional Recovery, Mental and Cognitive Health in Patients With Stroke
Brief Title: Motor Rehabilitation and Physical, Mental and Cognitive Health in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: *University of Jaén.
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: ACV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lokomat Group (Experimental): The intervention group will be composed of patients who have suffered a stroke and have alterations in mobility, balance and gait. These patients will be selected according to inclusion criteria such as clinical stability and ability to participate in a rehabilitation program. The group will receive structured physiotherapy sessions with a progressive approach to improve postural control, muscle strength, coordination and functional independence.
  Interventions: Other: Lokomat intervention

INTERVENTIONS:
Other: Lokomat intervention — The intervention will consist of an 8-week motor rehabilitation program, with 3 weekly sessions of 60 minutes each. In the first weeks, joint mobilization and postural control in a sitting position will be worked on, followed by muscle strengthening and balance re-education in a standing position. Subsequently, coordination exercises and assisted walking on different surfaces will be incorporated. In the final phase, independent walking and the integration of functional movements in daily life activities will be encouraged. The program will be adapted to the individual needs of each patient to optimize recovery and improve quality of life.

SUMMARY:
This study analyzes the effectiveness of a motor rehabilitation program in the functional recovery of stroke patients and its impact physiotherapy, occupational therapy, and neuropsychology are used to measure improvements in balance, mobility, independence in daily activities, and cognitive functions. The intervention involves the use of the Lokomat, a technologically advanced robot-assisted gait training device. Patients are supported in a harness on a treadmill while the robotic system guides their legs through a natural gait cycle. The results will help clarify the relationship between motor recovery and overall well-being, providing evidence to optimize therapeutic strategies for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ischemic or hemorrhagic stroke.
* Age equal to or greater than 18 years.
* Patients in the subacute or chronic phase of stroke (≥ 3 months since the event).
* Ability to participate in a motor rehabilitation program.
* Absence of advanced neurodegenerative diseases that may interfere with the evaluation of results.
* Ability to understand and follow basic instructions of the rehabilitation program.
* Informed consent signed by the patient or his/her legal representative.

Exclusion Criteria:

* People under 60 years of age.
* Presence of serious comorbidities that prevent physical activity or rehabilitation (e.g. severe heart failure, advanced chronic obstructive pulmonary disease).
* Patients with severe cognitive impairments that make it difficult to follow the program (e.g. advanced dementia).
* Use of drugs that significantly affect motor and cognitive function, interfering with the evaluation of rehabilitation.
* Presence of active infections or unstable medical conditions requiring hospitalization.
* History of another neurological disorder that may affect functional recovery (e.g. Parkinson's disease, multiple sclerosis).
* Participation in another rehabilitation program at the same time, which may interfere with the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Balance | Up to twelve weeks
  The Berg Scale is a widely used tool for assessing static and dynamic balance in adults with neuromotor impairments. It consists of 14 items that assess various functional tasks, such as standing, transferring, trunk rotation, and turning gait. Each item is scored on an ordinal scale from 0 to 4, with 0 indicating the lowest functional capacity and 4 indicating independent and safe performance of the task, with a maximum total score of 56 points. Scores below 45 are associated with an increased risk of falls. This scale has demonstrated high interobserver reliability (ICC > 0.95) and concurrent validity in stroke patients.
Postural Control | Up to twelve weeks
  The Postural Assessment Scale for Stroke Patients (PASS) is specifically designed to assess postural control in stroke patients, both in the acute and chronic phases. It includes 12 items that assess postural maintenance and changes in different positions (recumbent, sitting, and standing). Each item is scored from 0 to 3, with a maximum total score of 36 points. The PASS is particularly sensitive for detecting small functional changes during the early stages of post-stroke recovery and has demonstrated good discriminative and predictive validity for the evolution of postural control and gait. Its use is recom-mended for monitoring clinical progress in the rehabilitation setting.
Functional Independence | Up to twelve weeks
  The Barthel Index is a commonly used instrument for measuring functional inde-pendence in basic activities of daily living (BADL). It assesses a patient's ability to perform 10 activities, including feeding, dressing, toileting, mobility, and climbing and descending stairs, among others. Scoring varies by task, with a maximum of 100 points awarded, with higher scores indicating greater autonomy. The BI is sensitive to clinical changes after rehabilitation interventions and has high reliability (α > 0.90). It is widely used in clinical research with neurological populations, including post-stroke patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Agustín Aibar Almazán, Jaén, Spain